CLINICAL TRIAL: NCT05499962
Title: PrEP Initiation and Adherence Among Black SMM: A Social Network-Level Intervention
Brief Title: SNS and PrEP Initiation and Adherence in Black SMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Us Helping Us, People Into Living, Inc. (Other)
Responsible Party: Principal Investigator, DeMarc A. Hickson, PhD, Executive Director, Us Helping Us, People Into Living, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-USHE-104
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Recruit 30 PrEP-using Black SMM, including those who use substances, as Recruiters to identify and refer Network Associates to PrEP services. The pilot will occur in six blocks of up to 5 Recruiters to further develop all intervention procedures and enhance the SNS intervention's feasibility and acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP-using Black SMM as Recruiters (Other): Recruit 30 PrEP-using Black SMM, including those who use substances, as Recruiters to identify and refer Network Associates to PrEP services. The pilot will occur in six blocks of up to 5 Recruiters to further develop all intervention procedures and enhance the SNS intervention's feasibility and acceptability.
  Interventions: Behavioral: Social Networking Strategies

INTERVENTIONS:
Behavioral: Social Networking Strategies — Assess whether PrEP-using Black SMM can serve as an Interventionist to get their social and sexual network members to uptake and adhere to PrEP

SUMMARY:
Specific Aim 1. Conduct 18 focus groups among Black gay, bisexual and other sexual minority men (SMM; n=72-90) in the Washington, DC area of different age groups (18-24, 25-34, 35+) and various pre-exposure prophylaxis (PrEP) use profiles (i.e., PrEP naïve, current PrEP users, and discontinued PrEP; two per age-group and PrEP use profile) to understand intervention feasibility, acceptability and appropriateness, how the intervention can address experienced and perceived socio-structural barriers, and increase PrEP initiation and adherence among Black SMM in the Washington, District of Columbia (DC) area.

Specific Aim 2. Implement an iterative open-phase pilot of an SNS intervention to increase PrEP initiation among human immunodeficiency virus (HIV)-negative Black SMM, aged 18 years and above, in the Washington, DC area. Recruit 30 PrEP-using Black SMM, including those who use substances, as Recruiters to identify and refer Network Associates to PrEP services. The pilot will occur in six blocks of up to 5 Recruiters to further develop all intervention procedures and enhance the social networking strategy (SNS) intervention's feasibility and acceptability.

DETAILED DESCRIPTION:
The first 12 months (Phase 1: Formative Research) will be an intervention development/adaptation phase. Using a community-based participatory approach (n=18 age- and PrEP use profile-specific focus groups, of at least 4-5 participants each, totaling 72-90), participants will be asked about the social network dynamics and characteristics (e.g., influential network members, communication about PrEP as an HIV prevention method) that influenced their decision to initiate PrEP. Among participants with no PrEP use, they will be asked about the acceptability and feasibility of talking with PrEP-using Black SMM within their respective social network to support initiation along with preferences for relevant PrEP-related information from peers.

The following 12 months (Phase 2: Open-phase Pilot Study) will involve conducting an open pilot of the SNS intervention, in up to six batches of up to 5 participants (n=30), allowing for further intervention refinement. This will allow us to demonstrate participant feasibility and acceptance, which includes the ability to recruit network members, feasibility of intervention delivery, and changes in participant behaviors. It will allow for further evaluation of the feasibility of all study procedures, and refinement of intervention manual. Therefore, the expected outcome is a culturally relevant SNS intervention to increase PrEP initiation among Black SMM through PrEP-using social network members.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above
* Black or African American race
* Cisgender male identity
* Gay, bisexual or a male who has sex with other males
* Residence in the greater Washington, DC area (includes District of Columbia, Prince George's County, MD and Montgomery County, MD)
* Current PrEP use
* Confirmed HIV-negative status.

Exclusion Criteria:

* Being younger than 18 years of age ;
* Cisgender or transgender female identity
* Males having sex with women exclusively
* Being unable to speak or read English
* Reside outside of the defined greater Washington, DC area
* Being unable or unwilling to provide written informed consent
* Being unable to comply with the requirements of the protocol (e.g. persons with mental health conditions, persons who are intoxicated or incoherent for other reasons)
* Being a member of other vulnerable populations: pregnant women, children or wards of the state.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Black gay, bisexual and other sexual minority men (SMM)
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention as measured by Weiner et al., 2017. | During the peer-based debriefing sessions that occurs before a Recruiter is dismissed from the open-phase pilot.
  Assess the feasibility of intervention delivery method (i.e., PrEP-using SMM as the Interventionist/Recruiter).
Acceptability of Intervention as measured by Weiner et al., 2017. | During the peer-based debriefing sessions that occurs before a Recruiter is dismissed from the open-phase pilot.
  Assess the feasibility of intervention delivery method (i.e., PrEP-using SMM as the Interventionist/Recruiter).

SECONDARY OUTCOMES:
Recruited Network Members | Immediately after PrEP-using SMM enroll as an Interventionist (i.e., Recruiter)
  Proportion of Recruiters who recruit Network Associates
Network members on PrEP | Immediately after PrEP-using SMM enroll as an Interventionist (i.e., Recruiter)
  Number of Network Associates recruited
Comfortability of the Intervention as measured by an adaptation of Weiner et al., 2017. | During the peer-based debriefing sessions that occurs before a Recruiter is dismissed from the open-phase pilot.
  Extent to which Network Associates were comfortable with the intervention modality

CONTACTS AND LOCATIONS:
Overall Officials: DeMarc A Hickson, PhD, Principal Investigator — Executive Director
Locations (1):
- Us Helping Us, People Into Living, Inc., Washington D.C., District of Columbia, United States